CLINICAL TRIAL: NCT03267238
Title: Fecal Microbial Transplantation in Patients With Crohn's Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Ellen Li, Professor, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 973349
Record Dates: First submitted 2017-07-24; First posted 2017-08-30 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fecal Microbial transplantation (Experimental): Fecal Microbial Transplantation will be offered to patients eligible to be part of the study.
  Interventions: Biological: Fecal Microbial Transplantation

INTERVENTIONS:
Biological: Fecal Microbial Transplantation — Fecal Microbial Transplantation via will be offered to eligible Crohn's patient
  Other Names: FMT

SUMMARY:
Fecal Microbiota Transplantation will be offered to eligible Crohn's disease patient as Investigational New Drug treatment

DETAILED DESCRIPTION:
The following hypothesis will be tested in this study:

1. Fecal microbiota transplantation is a safe, tolerable procedure.
2. The fecal microbial diversity, composition and function in stool recipients after fecal transplantation will change to a similar microbial diversity, composition and functionality as found in donor stool.

Primary objectives:

1. To determine the short term safety and tolerability of fecal microbiota transplantation up to 12 weeks post-transplant in patients with Crohn's disease.

Secondary objectives:

1. To determine the long term safety and tolerability of fecal microbiota transplantation (FMT) up to one year post transplant in patients with Crohn's disease.
2. To compare microbial diversity in healthy donor stools compared to pre-FMT recipient stools collected from patients (recipients) with Crohn's disease.
3. To compare microbial composition in healthy donor stools compared to pre-FMT recipient stools from patients (recipients) with Crohn's disease.
4. To compare microbial function in healthy donor stools compared to pre-FMT recipient stools from patients (recipients) with Crohn's disease
5. To compare microbial diversity in healthy donor stools and pre-FMT recipient stools with 1 week post-transplant recipient stool samples collected from patients (recipients) with Crohn's disease.
6. To compare microbial composition in healthy donor stools and pre-FMT recipient stools with 1 week post-transplant recipient stool samples collected from patients (recipients) with Crohn's disease.
7. To compare microbial function in healthy donor stools and pre-FMT recipient stools with 1 week post-transplant recipient stool samples collected from patients (recipients) with Crohn's disease.
8. To compare microbial diversity in healthy donor stools and pre-FMT recipient stools with 12 week post transplant recipient stool samples collected from patients (recipients) with Crohn's disease.
9. To compare microbial composition in healthy donor stools and pre-FMT recipient stools with 12 week post transplant recipient stool samples collected from patients (recipients) with Crohn's disease.
10. To compare microbial function in healthy donor stools and pre-FMT recipient stools with 12 week post transplant recipient stool samples collected from patients (recipients) with Crohn's disease.
11. Stool calprotectin levels will be measured in the recipient at baseline pre-FMT, 1 week and 12 weeks post FMT to determine if FMT causes a statistically significant change.

ELIGIBILITY:
Inclusion Criteria for initial Fecal Microbial Transplant for Crohn's disease:

All patients age ≥7 years of age with established diagnosis of Crohn's disease made by a primary gastroenterologist based on history, physical examination, laboratory/radiological studies, and gastrointestinal histology, with one or more of the following criteria:

1. has been treated with steroid therapy for at least a month
2. has been treated with immunomodulatory therapy for at least a month
3. has been treated with biological therapy for at leaset a month

All patients or legal guardians of patients less than 18 years of age will have to give consent. The consent form will outline that although fecal microbiota transplantation appears safe based on past studies, a theoretical risk of transmission of an unrecognized infectious agent or substance exists and could result in an unexpected disease. All patients aged ≥7 and <18 years will have to give assent

Exclusion Criteria:

1. Patients less than 7 years of age
2. Scheduled for abdominal surgery within the next 12 weeks
3. Major abdominal surgery within the past 3 months
4. Pregnancy (This will be checked through a urine test on the day of procedure)
5. Anemia: Hemoglobin < 6 g/dL,
6. Neutropenia: Absolute Neutrophil Count <1500 Both of the above criteria will be checked via screening test or blood test reports within one month prior to the procedure
7. A known diagnosis of graft vs. host disease
8. Presence of an intra-abdominal or perianal abscess.
9. Presence of intestinal cutaneous fistula
10. Presence of severe intestinal stricture and/or intestinal obstruction
11. Administration of any investigational drug within the past 2 months
12. Use of a TNF-α antagonist within 2 weeks of the proposed date of transplantation
13. Bacteremia within past 4 weeks (28 days)
14. Severe Crohn's Disease, determined by Pediatric Crohns Disease Activity Index (PCDAI) value of more than 29.
15. Individuals with severe prior allergic reaction to food;
16. Individuals with intercurrent illness including but not necessarily limited to: febrile illness, decompensated liver cirrhosis, HIV/AIDS BMT within past 150 days, malignancy, or other severe immunodeficiency.
17. Individuals at increased risk for complications of endoscopy or procedural sedation (e.g., ASA classification IV and above).
18. Previous FMT

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 5 years
  Number of participants with treatment-related adverse events with grade greater than 2 within one year after FMT will be reported.

SECONDARY OUTCOMES:
To measure the effect of fecal microbial transplantation on microbial diversity in healthy donor stools compared to pre-FMT, 1 week post FMT, and 12 weeks post-FMT recipient stools. | 6 years
  Fecal DNA samples will undergo V3-V4 16S rRNA sequencing. Operational taxonomic units (OTUs) will be produced by clustering sequences with identical taxonomic assignments. Alpha diversity indices (e.g. Chao1, Shannon complexity H, Shannon Evenness H/Hmax) will be calculated inferred through 1000 replicate resamplings using Explicet. Beta diversity (Bray-Curtis and Jaccard distances) will be calculated for the recipient Pre-FMT, 1 week post-FMT and 12 weeks post-FMT as compared to their pared donor using the adonis function in the R vegan package at the phyla, family and genus level. A linear mixed model will be used to compare alpha-diversity (ShannonH) and beta-diversity (Bray-Curtis and Jaccard distance) between each timepoint (FMT) and each disease group (Group). P-values less than 0.05 were considered as statistically significant.
To measure the effect of fecal microbial transplantation on microbial composition in healthy donor stools compared to pre-FMT, 1 week post FMT, and 12 weeks post-FMT recipient stools. | 6 years
  Fecal DNA samples will undergo V3-V4 16S rRNA sequencing. . Operational taxonomic units (OTUs) will be produced by clustering sequences with identical taxonomic assignments. Linear mixed models analyses on individual OTUs at the genus level will be conducted on 105 OTUs after eliminating OTUs with an average relative abundance of < 0.001% in the donor and recipient pre-FMT samples, and after discarding OTUs where more than 75% of the samples had a zero count. To compare the relative abundance of each OTU between timepoints before and after FMT [pre-transplant recipient, 1-wk. post-FMT recipient, 3-mos. post-FMT recipient] and each disease group, a generalized linear mixed model (GLMM) or generalized estimating equation (GEE) will be used by taking the actual counts of each OTU as the outcomes that were assumed to follow a negative binomial distribution. The p-values will be adjusted for multiple comparisons by the Bonferroni correction or by the Benjamin-Hochberg method (FDR < 0.05).
To measure the effect of fecal microbial transplantation on microbial function using shotgun DNA metagenomic in healthy donor stools compared to pre-FMT, 1 week post FMT, and 12 weeks post-FMT recipient stools. | 6 years
  Fecal DNA samples will undergo shotgun DNA metagenomics sequencing. After removing human sequences, the Reads per kilobase gene length (RKP) will be calculated using HUMANN2 software for individual bacterial proteins/enzymes and pathways. . A linear mixed model will be used to compare RPK associated with pathways and individual proteins between each timepoint (FMT) and each disease group (Group). P-values less than 0.05 were considered as statistically significant.Linear mixed models analyses on the RPK associated with individual genes and pathways will be analyzed using linear mixed models between timepoints before and after FMT [pre-transplant recipient, 1-wk. post-FMT recipient, 3-mos. post-FMT recipient] and each disease group, a generalized linear mixed model (GLMM) or generalized estimating equation (GEE) were used by taking the actual RPK as the outcomes that will be assumed to follow a negative binomial distribution.
To measure the effect of fecal microbial transplantation on microbial function using bacterial metatranscriptomic sequencing | 6 years
  Fecal RNA samples will undergo bacterial metatranscriptomic RNA sequencing. After removing human sequences, the Reads per kilobase transcript (RKP) will be calculated for individual bacterial proteins/enzymes and pathways. A linear mixed model will be used to compare RPK associated with pathways and individual proteins between each timepoint (FMT) and each disease group (Group). P-values less than 0.05 were considered as statistically significant.
To measure the effect of fecal microbial transplantation on microbial function using targeted metabolomic assays. | 6 years
  Fecal samples will undergo extraction for targeted metabolomics analysis of short chain fatty acids (micrograms/gram stool) using gas chromatography-mass spectrometry, and of bile acids (microgram/gram stool) using liquid chromatography-mass spectrometry. A linear mixed model will be used to compare respectively short chain fatty acid and bile acid metabolites between each timepoint (FMT) and each disease group (Group). P-values less than 0.05 were considered as statistically significant.
Determine if FMT causes a statistically significant change in recipient fecal calprotectin levels | 6 years
  Fecal calprotectin (microgram/gram stool) levels will be measured as in the recipient at baseline pre-FMT, 1 week, and 12 weeks post FMT. A linear mixed model will be used to compare fecal calprotectin levels between each timepoint (FMT) and each disease group (Group). P-values less than 0.05 were considered as statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Li, MD, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT03267238/Prot_ICF_002.pdf